CLINICAL TRIAL: NCT00057538
Title: Curb, Alter, Lower, or Manage Stress in HIV: CALMS-HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: R21AT001159-01A1 (NIH)
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections
Keywords: HIV; Randomized Trial; Stress; Spirituality; Quality of Life; Complementary Therapies
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: Mantram Repetition

SUMMARY:
The purpose of this study is to determine the effectiveness of a stress management group intervention for people with HIV. The study will evaluate several outcomes, including perceived stress, quality of life, psychosocial factors, and physiological measures of stress.

DETAILED DESCRIPTION:
It is well documented that living with HIV/AIDS can cause a great amount of stress, and evidence suggests that stress may hasten HIV disease progression by increasing viral replication and suppressing the immune response. Stress management intervention studies using more complex combinations of cognitive and relaxation therapies have shown improvements in both psychological and physiological measures in HIV infected persons. However, no studies have focused on only one intervention or have addressed the spiritual component using a comparable control group to determine which of these interventions is most effective.

Participants will be randomly assigned to receive either a spiritually-based cognitive intervention to an educational control group. The intervention will be given over a 10-week period, with 5 weekly classes, 4 weekly automated phone calls, and one final class meeting. Assessments will be conducted at pre-intervention, fifth class midpoint, tenth week post-intervention, and 3-month follow-up. Time commitment can vary from 6 months to 9 months, depending on when participants are screened.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected for at least 6 months
* Ability to read and write English

Exclusion Criteria:

* Drug use within the past 6 months
* Cognitive impairment or dementia
* Diagnosis that may affect cortisol levels, such as diabetes, cancer, or asthma
* Loss of family/loved one in past 3 months
* Started a relaxation therapy in past 3 months
* History or current practice of the RISE program, rosary, chanting, or Transcendental Meditation (TM)
* Acute infection in past month
* Change of HAART or drug regimen in past month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-05; Study Completion 2003-05

PRIMARY OUTCOMES:
Intrusive Thoughts
Perceived Stress
Trait Anxiety
Trait Anger

SECONDARY OUTCOMES:
Spiritual Well-Being (FACIT-SpEx)
Quality of Life Enjoyment and Satisfaction
Ways of Coping
Urinary cortisol levels
Urinary catecholamines
Salivary cortisol levels

CONTACTS AND LOCATIONS:
Overall Officials: Jill E. Bormann, PhD, RN, Principal Investigator — California San Diego Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Background] Bormann, JE. Frequent, silent mantram repetition: A jacuzzi for the mind. Topics in Emergency Medicine 27(2): 163-166, 2005.